CLINICAL TRIAL: NCT05244577
Title: A Phase III Randomized, Double-blind, Placebo-controlled, Cross-over Study to Evaluate Olanzapine Combined With Fosaprepitant, Ondansetron, and Dexamethasone for Preventing Nausea and Vomiting in Patients With Testicular Cancer Receiving 5-day Cisplatin Combination Chemotherapy
Brief Title: Olanzapine Combined With Fosaprepitant, Ondansetron, and Dexamethasone for Preventing Nausea and Vomiting in Patients With Testicular Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shi Yanxia (Other)
Responsible Party: Sponsor-Investigator, Shi Yanxia, Principal Investigator, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-FXY-268
Record Dates: First submitted 2022-01-09; First posted 2022-02-17 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Olanzapine; CINV; Testicular Cancer by AJCC V6 and V7 Stage; Cisplatin
Keywords: testicular cancer; olanzapine; Cisplatin 5-day regimen; Nausea and vomiting
MeSH Terms: conditions — Testicular Neoplasms; Nausea; Vomiting | interventions — Olanzapine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olanzapine (Experimental): Ondansetron 8mg IV, D1-5 30 minutes before chemotherapy; Dexamethasone 6mg Po QD, D1-7; Fosaprepitant 150mg IVD D1,4, 60 minutes before chemotherapy; Olanzapine 5mg Po D1-7
  Interventions: Drug: Olanzapine Tablets
- Placebo (Placebo Comparator): Ondansetron 8mg IV, D1-5 30 minutes before chemotherapy; Dexamethasone 6mg Po QD, D1-7; Fosaprepitant 150mg IVD D1,4, 60 minutes before chemotherapy; Placebo 5mg Po D1-7
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olanzapine Tablets — Olanzapine,Ondansetron,Dexamethasone,Fosaprepitant
  Other Names: Olanzapine
  Arms: Olanzapine
Drug: Placebo — Placebo,Ondansetron,Dexamethasone,Fosaprepitant
  Arms: Placebo

SUMMARY:
This study aims to investigate the efficacy and safety of olanzapine combined with fosaprepitant, ondansetron and dexamethasone compared with placebo combined with fosaprepitant, ondansetron and dexamethasone in the prevention of nausea and vomiting in germ-cell tumors receiving 5-day cisplatin chemotherapy

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled, cross-over Phase III clinical study.

A total of 75 patients were enrolled in two sequential treatment groups (olanzapine-placebo and placebo-Olanzapine).

(1) The screening process begins after the patient signs the written informed consent. (2) Patients were randomly divided into control group (placebo) and experimental group (olanzapine). (3) Patients' effectiveness from the beginning of chemotherapy drug infusion (0 h on day 1) to day 10 (approximately 240 h) was monitored by patients' diary from 2 to 10 days after chemotherapy, in which patients should report episodes of vomiting in the previous 24 hours, use of remedial therapy, and assessment of daily nausea. Any episodes of vomiting or retching, as well as the time and date of use of rescue medications, should also be recorded. At days 2 to 6, patients were assessed on the visual analog scale (VAS) for the previous 24 hours. (4) The Hospital Anxiety and Depression Scale (HADS),and Life Index - Vomiting (FLIE) questionnaire of days 1-10 should be completed immediately after the log is completed on day 10. (5) During the study period, patients may receive "remedial treatment" for nausea or vomiting, and patients requiring remedial treatment are considered to have failed treatment because the primary endpoint is complete remission. However, patients receiving remedial treatment must continue to receive the study drug and complete the diary as directed.

ELIGIBILITY:
Inclusion Criteria

Patients must meet the following criteria for inclusion:

1. Pathology confirmed germ cell tumor (both spermatogonoma and non-spermatogonoma) and had no chemotherapy before;
2. Men;
3. Age ≥16 years old;
4. ECOG score of physical status 0-2;
5. Chemotherapy regimen containing 5-day cisplatin (20mg/m2, 100mg total;
6. No other nausea, vomiting, or use of any antiemetics within 72 hours prior to enrollment;
7. There are no clear brain metastases or other reasons for long-term systemic use of hormones;
8. The general condition is good, and the blood, liver and kidney functions meet the following standards:

   Hemoglobin: 90 g/L and above White blood cell count: 3.5 * 109 / L - 10.0 *109 / L Neutrophil count: 1.5* 109/L or above Platelet count: 90* 109/L or above Serum total bilirubin: below 1.5 times the upper limit of normal Serum AST, ALT and ALP: the upper limit of normal is below 2.5 times when the patient is present
9. Ability to read, understand and complete research questionnaires and journals, including visual analog scale (VAS);
10. Understand the study procedure and sign the informed consent in person to participate in the study

Exclusion Criteria

Patients who meet any of the following criteria will be excluded:

1. Digestive tract obstruction, water and electrolyte disorder;
2. Have central nervous system diseases (such as primary brain tumors, uncontrolled seizures, any history of brain metastases or strokes);
3. Contraindications to the use of glucocorticoids: ① Viral, bacterial, fungal and other infections that cannot be controlled by antibiotics;② Active gastric or duodenal ulcer;③ Severe hypertension, arteriosclerosis, diabetes; ④ Osteoporosis;⑤ Corneal ulcer;⑥Trauma or surgical repair period, fracture; ⑦Adeno-cortical hyperfunction; ⑧Severe mental illness and epilepsy; ⑨ patients with cardiac or renal dysfunction;
4. Patients with mental disabilities or severe emotional or mental disorders are considered unsuitable for inclusion in the study;
5. In addition to malignancy, the patient has an active infection (e.g. pneumonia, hepatitis) or any uncontrolled infection diseases (such as diabetic ketoacidosis), and the researchers believe may contribute to the study's findings confounding, or exposing patients receiving study drugs to unnecessary risks;
6. The patient is currently using any prohibited drugs, including medicinal marijuana or is currently using alcohol (Chinese Diagnostic criteria for drug dependence);
7. The patient received an unapproved (experimental) drug treatment within the past 4 weeks;
8. Taking oral olanzapine or other psychotropic drugs;
9. A history of hypersensitivity to fosappitan, 5-HT3 receptor antagonists or dexamethasone;
10. The patient cannot swallow the drugs;
11. The principal investigator considered the patients unsuitable for the study;
12. Inability or unwillingness to adhere to research protocols

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Complete Response From 0 to 240 Hours After Initiation chemotherapy | 1 to 10 days
  Complete Response was defined as no vomiting and no use of rescue medication

SECONDARY OUTCOMES:
Percentage of Participants With minimal nausea | 1-10 days
  Minimal nausea was defined as <25 mm on a visual analog scale
Percentage of Participants with total control | 1 to 10 days
  total control was defined as no vomiting, no rescue antiemetics, and no nausea
Severity of nausea | 1 to 10 days
Number of rescue medications | 1 to 10 days
  Number of rescue medications for nause and vormitting
Time to Treatment Failure in each group of participates | 1 to 10 days
  Time to treatment failure was defined as time to 1st emetic episode or use of rescue medication
Patient's satisfaction with anti-emetic therapy | 1 to 10 days
  The patient was asked to evaluate his satisfaction with the control of nausea and vomiting by recording two scales: Hospital Anxiety and Depression Scale and The Functional Living Index-Emesis questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Shi, PHD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Goding Sauer A, Fedewa SA, Butterly LF, Anderson JC, Cercek A, Smith RA, Jemal A. Colorectal cancer statistics, 2020. CA Cancer J Clin. 2020 May;70(3):145-164. doi: 10.3322/caac.21601. Epub 2020 Mar 5. PMID 32133645
- [Background] Herman TS, Einhorn LH, Jones SE, Nagy C, Chester AB, Dean JC, Furnas B, Williams SD, Leigh SA, Dorr RT, Moon TE. Superiority of nabilone over prochlorperazine as an antiemetic in patients receiving cancer chemotherapy. N Engl J Med. 1979 Jun 7;300(23):1295-7. doi: 10.1056/NEJM197906073002302. PMID 375088
- [Background] Hesketh PJ, Grunberg SM, Gralla RJ, Warr DG, Roila F, de Wit R, Chawla SP, Carides AD, Ianus J, Elmer ME, Evans JK, Beck K, Reines S, Horgan KJ; Aprepitant Protocol 052 Study Group. The oral neurokinin-1 antagonist aprepitant for the prevention of chemotherapy-induced nausea and vomiting: a multinational, randomized, double-blind, placebo-controlled trial in patients receiving high-dose cisplatin--the Aprepitant Protocol 052 Study Group. J Clin Oncol. 2003 Nov 15;21(22):4112-9. doi: 10.1200/JCO.2003.01.095. Epub 2003 Oct 14. PMID 14559886
- [Background] Schmoll HJ, Aapro MS, Poli-Bigelli S, Kim HK, Park K, Jordan K, von Pawel J, Giezek H, Ahmed T, Chan CY. Comparison of an aprepitant regimen with a multiple-day ondansetron regimen, both with dexamethasone, for antiemetic efficacy in high-dose cisplatin treatment. Ann Oncol. 2006 Jun;17(6):1000-6. doi: 10.1093/annonc/mdl019. Epub 2006 Mar 8. PMID 16524979
- [Background] Albany C, Brames MJ, Fausel C, Johnson CS, Picus J, Einhorn LH. Randomized, double-blind, placebo-controlled, phase III cross-over study evaluating the oral neurokinin-1 antagonist aprepitant in combination with a 5HT3 receptor antagonist and dexamethasone in patients with germ cell tumors receiving 5-day cisplatin combination chemotherapy regimens: a hoosier oncology group study. J Clin Oncol. 2012 Nov 10;30(32):3998-4003. doi: 10.1200/JCO.2011.39.5558. Epub 2012 Aug 20. PMID 22915652
- [Background] Ioroi T, Furukawa J, Kume M, Hirata S, Utsubo Y, Mizuta N, Miyake H, Fujisawa M, Hirai M. Phase II study of palonosetron, aprepitant and dexamethasone to prevent nausea and vomiting induced by multiple-day emetogenic chemotherapy. Support Care Cancer. 2018 May;26(5):1419-1423. doi: 10.1007/s00520-017-3967-2. Epub 2017 Nov 16. PMID 29147855
- [Background] Olver IN, Grimison P, Chatfield M, Stockler MR, Toner GC, Gebski V, Harrup R, Underhill C, Kichenadasse G, Singhal N, Davis ID, Boland A, McDonald A, Thomson D; Australian and New Zealand Urogenital and Prostate Cancer Trials Group. Results of a 7-day aprepitant schedule for the prevention of nausea and vomiting in 5-day cisplatin-based germ cell tumor chemotherapy. Support Care Cancer. 2013 Jun;21(6):1561-8. doi: 10.1007/s00520-012-1696-0. Epub 2012 Dec 30. PMID 23274926
- [Background] Grunberg S, Chua D, Maru A, Dinis J, DeVandry S, Boice JA, Hardwick JS, Beckford E, Taylor A, Carides A, Roila F, Herrstedt J. Single-dose fosaprepitant for the prevention of chemotherapy-induced nausea and vomiting associated with cisplatin therapy: randomized, double-blind study protocol--EASE. J Clin Oncol. 2011 Apr 10;29(11):1495-501. doi: 10.1200/JCO.2010.31.7859. Epub 2011 Mar 7. PMID 21383291
- [Background] Hashimoto H, Abe M, Tokuyama O, Mizutani H, Uchitomi Y, Yamaguchi T, Hoshina Y, Sakata Y, Takahashi TY, Nakashima K, Nakao M, Takei D, Zenda S, Mizukami K, Iwasa S, Sakurai M, Yamamoto N, Ohe Y. Olanzapine 5 mg plus standard antiemetic therapy for the prevention of chemotherapy-induced nausea and vomiting (J-FORCE): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2020 Feb;21(2):242-249. doi: 10.1016/S1470-2045(19)30678-3. Epub 2019 Dec 11. PMID 31838011

DOCUMENTS (2):
  • Study Protocol (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT05244577/Prot_000.pdf
  • Informed Consent Form (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT05244577/ICF_001.pdf